CLINICAL TRIAL: NCT03080311
Title: A Phase I Study of the Safety, Pharmacokinetic and Pharmacodynamic Properties of Intravenously Administered APG-1252 in Patients With Small Cell Lung Cancer (SCLC) or Other Solid Tumors
Brief Title: A Study of APG-1252 in Patients With SCLC or Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG-1252-US-001
Record Dates: First submitted 2017-02-12; First posted 2017-03-15 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Small Cell Lung Cancer; Solid Tumor
Keywords: Bcl-2/Bcl-xL dual inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pelcitoclax; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APG-1252 (Experimental): An accelerated dose escalation scheme will be utilized initially with one patient enrolled per cohort. If at 10 mg or 20 mg dose level, any occurrence in cycle 1 of one ≥ Grade 2 adverse event related or possibly related to APG-1252 (graded as per the National Cancer Institute's Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.0) is the trigger for converting to a standard 3+3 design at that dose level.
  Interventions: Drug: APG-1252

INTERVENTIONS:
Drug: APG-1252 — Multiple dose cohorts, 30 minute IV infusion, twice weekly for 3 weeks of a cycle with 28 days.
  Other Names: APG-1252 for injection

SUMMARY:
APG-1252 is a highly potent Bcl-2 family protein inhibitor, a promising drug candidate which shown high binding affinities to Bcl-2, Bcl-xL and Bcl-w. The preclinical studies have shown that APG-1252 alone achieves complete and persistent tumor regression in multiple tumor xenograft models with a twice weekly or weekly dose-schedule, including SCLC, colon, breast and acute lymphocytic leukemia (ALL) cancer xenografts; achieves strong synergy with the chemotherapeutic agents, indicating that APG-1252 may have a broad therapeutic potential for the treatment of human cancer as a single agent and in combination with other classes of anticancer drugs. APG-1252 is intended for the treatment of patients with SCLC or other solid tumors.

This is a multi-center, open-label, dose escalation Phase I study to determine the MTD and DLTs of intravenously administered APG-1252. After dose escalation to 240mg twice weekly, 2 dose cohorts two different dosing schedules including weekly and twice weekly will be assessed to evaluate for safety, tolerability, pharmacokinetics (PK) and preliminary anti-tumor efficacy. Treatment with APG-1252 will be administered to 30-60 patients at approximately 2 investigational sites in US.

DETAILED DESCRIPTION:
In dose cohort 1, patients will be treated in cycles, which are defined by APG-1252 intravenous administration on Days 1, 4, 8, 11, 15, 18 and 22, over a 28-day cycle the start dose is 10mg.

After dose escalation to 240mg twice weekly in dose cohort 1, dose cohort 2 will be performed with dose cohort 1 parallelly, patients will be treated in the same 28-day-cycles, APG-1252 intravenous administration on Days 1, 8, 15, and 22, the start dose is 240mg.

In both dose cohorts' patients could continue to receive cycles of APG-1252 until disease progress or unacceptable toxicity.

Study drug will be administered by intravenous infusion for 30 minutes at the investigational site by site staff.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed small cell lung cancer (SCLC) or other solid tumors
2. Male or non-pregnant, non-lactating female patients age ≥18 years
3. Locally advanced or metastatic disease for which no standard therapy is judged appropriate by the investigator
4. Eastern Cooperative Oncology Group (ECOG) Performance Status < 2
5. Adequate hematologic function as indicated by:

   1. Platelet count ≥ 100,000/mm˄3
   2. Hemoglobin ≥ 9.0g/dL Platelet count ≥ 100,000/mm˄3
   3. Absolute neutrophil count (ANC) ≥1000/µL
6. Adequate renal and liver function as indicated by:

   1. Serum creatinine ≤ 1.5 x upper limit of normal (ULN); if serum creatinine is >1.5 X ULN, creatinine clearance must be ≥ 50 mL/min
   2. Total bilirubin ≤1.5 x ULN; If Gilbert's Syndrome may have Bilirubin> 1.5 x ULN
   3. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤3 x ULN of institution's normal range; for patients with known liver metastases, AST and ALT may be ≤ 5 x ULN
   4. Coagulation: activated partial thromboplastin time (aPTT) and prothrombin time (PT)<1.2 x the upper limit of normal
7. Brain metastases with clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of CNS disease progression as determined by CT or MRI within 21 days prior to the first dose of study drug
8. Willingness to use contraception by a method that is deemed effective by the investigator by both males and female patients of child bearing potential (postmenopausal women must have been amenorrheal for at least 12 months to be considered of non-childbearing potential) and their partners throughout the treatment period and for at least three months following the last dose of study drug
9. Ability to understand and willingness to sign a written informed consent form
10. Willingness and ability to comply with study procedures and follow-up examination

Exclusion Criteria:

1. Receiving concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy, with the exception of hormones for hypothyroidism or estrogen replacement therapy (ERT), anti estrogen analogs, agonists required to suppress serum testosterone levels); or any investigational therapy, or has had tumor embolization or tumor lysis syndrome (TLS) within 14 days prior to the first dose of study drug
2. Steroid therapy for anti-neoplastic intent within 7 days prior to the first dose of study drug
3. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to < Grade 2
4. Known bleeding diathesis/disorder
5. Recent history of non-chemotherapy induced thrombocytopenia associated bleeding within 1 year prior to first dose of study drug
6. Have active immune thrombocytopenic purpura (ITP), active autoimmune hemolytic anemia (AIHA), or a history of being refractory to platelet transfusions (within 1 year prior to the first dose of study drug)
7. Serious gastrointestinal bleeding within 3 months
8. Use of therapeutic doses of anti-coagulants is excluded, along with anti-platelet agents; low-dose anticoagulation medications that are used to maintain the patency of a central intravenous catheter are permitted
9. Received a biologic (G-CSF, GM-CSF or erythropoietin) within 28 days prior to the first dose of study drug
10. Failure to recover adequately, as judged by the investigator, from prior surgical procedures. Patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry
11. Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry
12. Neurologic instability per clinical evaluation due to tumor involvement of the central nervous system (CNS). Patients with CNS tumors that have been treated, are asymptomatic and who have discontinued steroids (for the treatment of CNS tumors) for >28 days may be enrolled
13. Active symptomatic fungal, bacterial and/or viral infection including, but not limited to, active human immunodeficiency virus (HIV) or viral hepatitis (B or C)
14. Diagnosis of fever and neutropenia within 1 week prior to study drug administration
15. Uncontrolled concurrent illness including, but not limited to: serious uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements
16. Prior treatment with Bcl-2/Bcl-xL inhibitors
17. Any other condition or circumstance of that would, in the opinion of the investigator, make the patient unsuitable for participation in the study
18. Known clinically active hepatitis B or hepatitis C infection. Testing for hepatitis B and C is not required for study enrollment.
19. Known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) determination | 28 days
  Number of participants with APG-1252 treatment-related adverse events as assessed by NCI CTCAE v4.03
Maximum tolerated dose (MTD) determination | 18 - 24 months
  If ≥ 2/6 patients develop a DLT at any dose level, then this dose will be declared as the MTD

SECONDARY OUTCOMES:
Pharmacokinetic evaluation | 18 - 24 months
  Peak plasma concentration (Cmax) will be assessed on all participants with APG-1252 treatments
Pharmacokinetic evaluation | 18 - 24 months
  Area under the plasma concentration versus time curve (AUC) will be assessed on all participants with APG-1252 treatments
Pharmacodynamic evaluation | 18-24 months
  Platelet counts will be measured on the participants with APG-1252 treatments
Pharmacodynamic evaluation | 18-24 months
  Bcl-2 protein in peripheral blood mononuclear cells (PBMCs) will be measured on the participants with APG-1252 treatments
Pharmacodynamic evaluation | 18-24 months
  Activation of apoptosis will be measured on the participants with APG-1252 treatments
Preliminary efficacy assessment | 18-24 months
  Patients will be evaluated for response every 2 cycles (i.e., 8 weeks), according to the new response evaluation criteria in solid tumors: revised RECIST Guideline, Version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (2):
- United States (2):
  - START Midwest, Grand Rapids, Michigan
  - The START Center for Cancer Care, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No